CLINICAL TRIAL: NCT03028467
Title: A Phase 1/2, Double-Blind, Placebo-Controlled Study of the Pharmacokinetics, Safety and Tolerability of GSK3196165 in Combination With Methotrexate Therapy, in Japanese Subjects With Active Moderate-Severe Rheumatoid Arthritis Despite Treatment With Methotrexate
Brief Title: Evaluation of Pharmacokinetics and Safety of GSK3196165 in Combination With Methotrexate in Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201789
Record Dates: First submitted 2017-01-10; First posted 2017-01-23 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: GSK3196165; Active Rheumatoid Arthritis; Methotrexate; Monoclonal Antibody; Efficacy; Electrocardiogram; Tolerability; Pharmacokinetics; Japanese Subjects
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GSK3196165 Dose 1 (Experimental): Participants will receive GSK3196165 Dose 1 weekly as a single subcutaneous (SC) injection by an un-blinded administrator. There will be 5 weekly injections (Days 1, 8, 15, 22 and 29), then every other week (EOW) injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants will also receive a stable dose of methotrexate during the Treatment Period.
  Interventions: Drug: GSK3196165 Dose 1; Drug: Methotrexate; Drug: Folic acid
- GSK3196165 Dose 2 (Experimental): Participants will receive GSK3196165 Dose 2 weekly as a single SC injection by an un-blinded administrator. There will be 5 weekly injections (Days 1, 8, 15, 22 and 29), then EOW injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants will also receive a stable dose of methotrexate during the Treatment Period.
  Interventions: Drug: GSK3196165 Dose 2; Drug: Methotrexate; Drug: Folic acid
- GSK3196165 Dose 3 (Experimental): Participants will receive GSK3196165 Dose 3 weekly as a single SC injection by an un-blinded administrator. There will be 5 weekly injections (Days 1, 8, 15, 22 and 29), then EOW injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants will also receive a stable dose of methotrexate during the Treatment Period.
  Interventions: Drug: GSK3196165 Dose 3; Drug: Methotrexate; Drug: Folic acid
- Placebo (Placebo Comparator): Participants will receive placebo weekly as a single SC injection by an un-blinded administrator. There will be 5 weekly injections (Days 1, 8, 15, 22 and 29), then EOW injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants will also receive a stable dose of methotrexate during the Treatment Period.
  Interventions: Drug: Methotrexate; Drug: Placebo; Drug: Folic acid

INTERVENTIONS:
Drug: GSK3196165 Dose 1 — GSK3196165 is supplied as liquid and will be administered as SC injection.
  Arms: GSK3196165 Dose 1
Drug: GSK3196165 Dose 2 — GSK3196165 is supplied as liquid and will be administered as SC injection.
  Arms: GSK3196165 Dose 2
Drug: GSK3196165 Dose 3 — GSK3196165 is supplied as liquid and will be administered as SC injection.
  Arms: GSK3196165 Dose 3
Drug: Methotrexate — Methotrexate capsule/tablet 8-16 mg per week is given orally.
Drug: Placebo — Placebo is supplied as liquid as sterile 0.9% sodium chloride solution and will be administered as SC injection.
  Arms: Placebo
Drug: Folic acid — Folic acid tablet 5 mg per week is given orally.

SUMMARY:
This is a randomized, double-blind, parallel group, 3 dosage level, placebo-controlled, Phase 1/2 study designed to evaluate the pharmacokinetics, safety, tolerability, and efficacy of the monoclonal antibody GSK3196165, in Japanese subjects with active moderate-severe rheumatoid arthritis (RA) despite treatment with methotrexate(MTX). The subjects will receive GSK3196165 in combination with methotrexate therapy for the 12 weeks of treatment period. Approximately 55 subjects will be screened to achieve 40 randomized subjects, so as to have approximately 10 subjects in each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Age: >=20 years at the time of signing informed consent - Japanese rheumatoid arthritis (RA) subjects who meets American College of Rheumatology or European League Against Rheumatism (ACR/EULAR) 2010 RA Classification Criteria
* Functional class I, II or III defined by the 1992 ACR Classification of Functional Status in RA
* Disease duration of >=12 weeks (time from onset of subject-reported symptoms of either pain or stiffness or swelling in hands, feet or wrists).
* Swollen joint count of >=4 (66-joint count) and tender joint count of >=4 (68-joint count) at screening and at Day 1
* DAS28(CRP) >=3.2 at screening
* C-Reactive Protein (CRP) >=0.5 milligrams (mg)/deciliter (dL) at screening
* Must have previously received methotrexate (MTX) (8-16 mg weekly) orally for at least 12 weeks before screening, with a stable and tolerated dose for >=4 weeks prior to Day 1
* >=40 kilograms (kg) - Male or female subjects are eligible to participate so long as they meet and agree to abide by the contraceptive criteria
* Written informed consent prior to any of the screening procedures including discontinuation of prohibited medications
* Willing to continue or initiate treatment with oral folic acid (5 mg/week) and be treated during the entire study (mandatory co-medication for MTX treatment)
* Diffusing capacity of lung for carbon monoxide (DLCO) >=60% predicted; forced expiratory volume in 1 second (FEV1) >=70% predicted; forced vital capacity (FVC) >=80% predicted

  * For subjects with DLCO values ≥60% to <70%, a baseline chest high-resolution computed tomography (HRCT) must be performed during the screening period, and it is recommended that the subject be reviewed by a local pulmonologist to exclude significant pre-existing respiratory disease.
* No evidence of active or latent infection with Mycobacterium tuberculosis (TB), as defined by all of the following:

  * No history of active or latent TB infection irrespective of treatment status
  * A negative T-spot test within 4 weeks of baseline (Day 1)
  * Chest X-ray within 12 weeks of Day 1, locally read by a radiologist, with no evidence of current or previous pulmonary tuberculosis

Exclusion Criteria:

* Pregnant or lactating women
* History of other inflammatory rheumatologic or autoimmune disorders, other than Sjögren's syndrome secondary to RA
* History of any respiratory disease which (in the opinion of the investigator) would compromise subject safety or the ability of the subject to complete the study (e.g. significant interstitial lung disease, such as pulmonary fibrosis, chronic obstructive pulmonary disease (COPD), moderate-severe asthma, bronchiectasis, previous pulmonary alveolar proteinosis (PAP)
* Clinically-significant or unstable (in the opinion of the investigator) persistent cough or dyspnea that is unexplained
* QT interval corrected for heart rate (QTc) >450 milliseconds (msec) or QTc >480 msec for subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF)
* Liver function tests: alanine aminotransferase (ALT) >=1.5x upper limit of normal (ULN); aspartate transaminase (AST) >=1.5xULN; alkaline phosphatase and bilirubin >=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment)
* Clinically significant unstable or uncontrolled acute or chronic disease (e.g., cardiovascular including uncompensated congestive cardiac failure New York Heart Association [NYHA] III or IV, myocardial infarction within 12 months, unstable angina pectoris, uncontrolled hypertension, uncontrolled hypercholesterolemia) pulmonary, hematologic, gastrointestinal (including Crohn's Disease or ulcerative colitis), hepatic, renal, neurological, psychiatric, malignancy, endocrinological or infectious diseases, which, in the opinion of the investigator, could confound the results of the study or put the subject at undue risk
* A history of malignant neoplasm within the last 10 years or breast cancer within the last 20 years, except for non-melanoma skin cancers that have been excised and cured or carcinoma in situ of the uterine cervix
* Kidney disease: Current or history of renal disease, or estimated creatinine clearance <60 milliliter (mL)/minute (min)/1.73 m2 (MDRD formula) or serum creatinine >1.5xULN within 4 weeks of Day 1
* Hereditary or acquired immunodeficiency disorder, including immunoglobulin deficiency
* History of infected joint prosthesis at any time, with the prosthesis still in situ. History of leg ulcers, catheters, chronic sinusitis or recurrent chest or urinary tract infections
* Active infections, or history of recurrent infections (excluding recurrent fungal infections of the nail bed), or have required management of acute or chronic infections, as follows:

  * Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria)
  * OR Hospitalization for treatment of infection within 26 weeks of Day 1
  * OR Use of parenteral (Intravenous (IV) or Intramuscular (IM) antimicrobials (antibacterials, antivirals, antifungals, or antiparasitic agents) within 26 weeks of Day 1 or oral antimicrobials within 2 weeks of Day 1
* A vaccination (live or attenuated) within 30 days of Day 1 or Bacillus Calmette-Guérin (BCG) vaccination within 1 year of Day 1, or a live vaccination planned during the course of the study (including follow-up period).
* Any surgical procedure, including bone or joint surgery/synovectomy within 12 weeks prior to Day 1 or any planned surgery within the duration of the study (including follow-up period)
* Use of prohibited medications Prior to AND throughout the study:

Any conventional DMARDs other than MTX (including sulfasalazine, bucillamine, iguratimod, tacrolimus) should be withdrawn at least 2 weeks prior to Day 1.

Subjects may require longer to discontinue azathioprine or leflunomide prior to Day 1: Azathioprine must be discontinued >=4 weeks prior to randomization; Leflunomide must be discontinued >=12 weeks prior to Day 1 (or >=14 days after 11 days of standard cholestyramine or activated charcoal washout).

* For these subjects, written informed consent for the study must be obtained prior to beginning the screening period. However, other screening assessments, other than consent, must occur within 4 weeks prior to Day 1.
* Any biologic agents (such as Tumor necrosis factor (TNF) inhibitors [including adalimumab, etanercept, infliximab, certolizumab pegol, golimumab] or non-TNF inhibitors [including abatacept, rituximab, tocilizumab, belimumab]).
* Any Janus kinase (JAK) inhibitors (such as tofacitinib).
* Any anti-rheumatic investigational compounds.
* Any alkylating agents (such as cyclophosphamide).
* Plasmapheresis or intravenous immunoglobulin (IVIG) within 26 weeks of Day 1.

Corticosteroids:

* Any Intramascular (IM), Intravenous (IV) or Intra-arterial (IA) corticosteroids within 8 weeks of Day 1.
* Oral corticosteroids:

  * Any treatment with >10 mg/day dose oral prednisolone (or equivalent) within 4 weeks of Day 1.
  * New oral corticosteroid or changes in corticosteroid dose within the 4 weeks prior to Day 1. (New topical steroids and immunosuppressive agents (e.g., eye drops, creams) are permitted)
* Non-steroidal anti-inflammatory drugs (NSAIDs):

  * New or change in dose of NSAID within 2 weeks of Day 1
* Any non-anti-rheumatic investigational treatment must be discontinued for at least 4 weeks or 5 half-lives, whichever is longer, prior to Day 1
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within a year prior to Day 1
* History of sensitivity to any of the study treatments, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Abnormal chest X-ray within 12 weeks of Day 1 (locally read and reported by a radiologist) judged by the investigator as clinically-significant
* Any Grade 3 or 4 hematology or clinical chemistry laboratory abnormality, within 4 weeks of Day 1
* Hemoglobin ≤9 g/dL; white blood cell count ≤3.0 x 109/L; platelet count ≤100 x 109/L; absolute neutrophil count ≤1.5 x 109/L; lymphocyte count ≤0.5 x 109/L within 4 weeks of Day 1
* Serologic evidence of current/previous Hepatitis B virus (HBV) infection based on the results of testing for Hepatitis B surface antigen (HBsAg) and anti-Hepatitis B core (anti-HBc) antibody as follows within 4 weeks of Day 1

  * Subjects positive for HBsAg and/or positive for anti-HBc antibody (regardless of anti-HBs antibody status) are excluded
  * Subjects with positive anti-HBs antibody and HBV-DNA (>=2.1 log copies/mL) are excluded.
* Hepatitis C: Positive test for Hepatitis C virus (HCV) antibody confirmed on a subsequent blood sample by ribonucleic acid - polymerized chain reaction (RNA-PCR) assay within 4 weeks of Day 1.

  * Subjects who are positive for Hepatitis C antibody and negative when the Hepatitis C RNA-PCR assay is performed on a subsequent sample will be eligible to participate. Subjects who are positive for Hepatitis C antibody and have a positive result for the HCV when the Hepatitis C RNA-PCR assay is performed on the subsequent sample will not be eligible to participate
* Positive serology for human immunodeficiency virus (HIV) 1 or 2 (within 4 weeks of Day 1)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (9):
- Japan (9):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: SAP
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted to assess pharmacokinetics (PK), safety, tolerability and efficacy of GSK3196165 for 12 weeks, in combination with Methotrexate (MTX), in Japanese participants with active moderate-severe rheumatoid arthritis (RA) despite treatment with MTX. Participants were enrolled at 15 centers in Japan from 24-Jan-2017 to 30-Jun-2017.
Pre-assignment Details: A total of 35 participants were screened, and 20 participants failed screening because of not met eligibility criteria (18 participants) and withdrawal by participant (2 participants). Hence, a total of 15 participants were enrolled and randomized to study treatment.
Groups:
- Placebo: Participants received placebo weekly as a single subcutaneous (SC) injection by an un-blinded administrator. There were 5 weekly injections (Days 1, 8, 15, 22 and 29), then every other week (EOW) injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants also received a stable dose of MTX during the Treatment Period.
- GSK3196165 45 mg: Participants received GSK3196165 45 milligram (mg) weekly as a single SC injection by an un-blinded administrator. There were 5 weekly injections (Days 1, 8, 15, 22 and 29), then EOW injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants also received a stable dose of MTX during the Treatment Period.
- GSK3196165 90 mg: Participants received GSK3196165 90 mg weekly as a single SC injection by an un-blinded administrator. There were 5 weekly injections (Days 1, 8, 15, 22 and 29), then EOW injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants also received a stable dose of MTX during the Treatment Period.
- GSK3196165 180 mg: Participants received GSK3196165 180 mg weekly as a single SC injection by an un-blinded administrator. There were 5 weekly injections (Days 1, 8, 15, 22 and 29), then EOW injections at Days 43, 57 and 71 (Weeks 6, 8 and 10 respectively). Participants also received a stable dose of MTX during the Treatment Period.
Period: Overall Study
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Started | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg | Total
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (14.45) | 58.0 (15.72) | 66.5 (2.52) | 52.0 (9.20) | 57.1 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 3 | 9
  Male | 1 | 1 | 3 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Japanese/East Asian Heritage (EAH)/South EAH | 4 | 3 | 4 | 4 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK3196165
Description: Blood samples were collected at pre-dose on Days 1, 8, 15, 29, 57 and 71; and at any time during visit on Days 3, 74, 85, 106, 127 and 155. PK parameters were calculated by non-compartmental analysis using the concentration data after last dosing (Day 71). Only those participants whose parameters could be determined were analyzed. PK Population included all GSK3196165-treated participants from whom PK samples were collected and analyzed.
Time Frame: Pre-dose on Days 1, 8, 15, 29, 57 and 71; anytime during visit on Days 3, 74, 85, 106, 127 and 155
Population: PK Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Nanogram per milliliter (ng/mL)
Arm/Group | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 2 | 3 | 4
Nanogram per milliliter (ng/mL) | 699.92 [48.18 to 10167.77] | 1444.88 [148.02 to 14104.11] | 3924.10 [3375.18 to 4562.30]

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration (AUC [0-t]), AUC From Time Zero Extrapolated to Infinity (AUC [0-inf]), AUC Over the Dosing Interval (AUCtau) of GSK3196165
Description: Blood samples were collected at pre-dose on Days 1, 8, 15, 29, 57 and 71; and at any time during visit on Days 3, 74, 85, 106, 127 and 155. PK parameters were calculated by non-compartmental analysis using the concentration data after last dosing (Day 71). NA indicates data was not available as geometric mean and/or 95 percent confidence interval could not be calculated when number of participant was not sufficient.
Time Frame: Pre-dose on Days 1, 8, 15, 29, 57 and 71; anytime during visit on Days 3, 74, 85, 106, 127 and 155
Population: PK Population. Only those participants whose parameters could be determined were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*Nanogram per milliliter (hr*ng/mL)
Arm/Group | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 3 | 4 | 4
Hour*Nanogram per milliliter (hr*ng/mL)
  AUC (0-t), n=2, 3, 4: number analyzed (Participants) | 2 | 3 | 4
  AUC (0-t), n=2, 3, 4 | 189948.606 [508.091 to 71011815.710] | 386497.495 [32248.035 to 4632229.918] | 1186604.746 [589936.272 to 2386750.721]
  AUC (0-inf), n=0, 1, 2: number analyzed (Participants) | 0 | 1 | 2
  AUC (0-inf), n=0, 1, 2 |  | 732243.847 [NA to NA] — NA indicates data was not available as 95 percent confidence interval could not be calculated when number of participant was not sufficient. | 1097422.958 [106189.728 to 11341371.436]
  AUCtau, n=1, 3, 4: number analyzed (Participants) | 1 | 3 | 4
  AUCtau, n=1, 3, 4 | 196562.287 [NA to NA] — NA indicates data was not available as 95 percent confidence interval could not be calculated when number of participant was not sufficient. | 303167.467 [38999.824 to 2356690.471] | 787570.414 [570081.863 to 1088031.733]

3. Primary Outcome: Time to Reach Cmax (Tmax) of GSK3196165
Description: Blood samples were collected at pre-dose on Days 1, 8, 15, 29, 57 and 71; and at any time during visit on Days 3, 74, 85, 106, 127 and 155. PK parameters were calculated by non-compartmental analysis using the concentration data after last dosing (Day 71).
Time Frame: Pre-dose on Days 1, 8, 15, 29, 57 and 71; anytime during visit on Days 3, 74, 85, 106, 127 and 155
Population: PK Population. Only those participants whose parameters could be determined were analyzed.
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 2 | 3 | 4
Hour | 48.99167 [46.3500 to 51.6333] | 70.61667 [47.2500 to 94.0667] | 69.80000 [47.4000 to 70.8000]

4. Primary Outcome: Terminal Half-life (t1/2) of GSK3196165
Description: Blood samples were collected at pre-dose on Days 1, 8, 15, 29, 57 and 71; and at any time during visit on Days 3, 74, 85, 106, 127 and 155. PK parameters were calculated by standard non-compartmental analysis from the concentration data after last dosing (Day 71). NA indicates data was not available as 95 percent confidence interval could not be calculated when number of participant was not sufficient.
Time Frame: Pre-dose on Days 1, 8, 15, 29, 57 and 71; anytime during visit on Days 3, 74, 85, 106, 127 and 155.
Population: PK Population. Only those participants whose parameters could be determined were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 0 | 1 | 2
Hour |  | 282.85265 [NA to NA] — NA indicates data was not available as 95 percent confidence interval could not be calculated when number of participant was not sufficient. | 245.12966 [66.51778 to 903.34570]

5. Primary Outcome: Number of Participants With Any Adverse Event (AE), Serious AE (SAE) and Adverse Events of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. AESI included serious infections including serious respiratory infections and tuberculosis and opportunistic infections, neutropenia (grade 3 or 4), respiratory events, pulmonary alveolar proteinosis, hypersensitivity reactions including anaphylaxis and injection site reactions.
Time Frame: Up to 22 weeks
Population: Intent-to-Treat (ITT) Population. It included all participants who were randomized to treatment and who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants
  Any AE | 3 | 2 | 3 | 2
  Any SAE | 1 | 0 | 0 | 0
  Any AESI | 2 | 0 | 1 | 0

6. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital sign measurements including SBP and DBP were measured after 5 minutes rest before each reading. Baseline was considered as the latest pre-dose assessment. The change from Baseline is defined as the difference between the post-dose visit value and Baseline value.
Time Frame: Baseline and up to 22 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Millimeter of mercury
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Millimeter of mercury
  SBP, Week 1 | -0.3 (8.62) | -7.7 (2.89) | -15.0 (17.36) | -1.0 (8.45)
  SBP, Week 2 | -1.8 (8.34) | -6.7 (12.06) | -4.5 (12.48) | 1.5 (1.91)
  SBP, Week 3 | 0.5 (4.80) | -1.7 (12.01) | -10.5 (20.47) | -0.8 (6.02)
  SBP, Week 4 | -5.8 (10.14) | -11.3 (17.10) | -3.3 (17.88) | 6.3 (7.63)
  SBP, Week 6 | -2.0 (5.66) | -12.7 (11.59) | -1.3 (15.50) | -2.3 (11.62)
  SBP, Week 8 | -6.3 (7.41) | -3.0 (13.00) | -5.8 (18.55) | 3.8 (2.22)
  SBP, Week 10 | 2.3 (4.86) | 6.7 (5.03) | -11.8 (23.04) | -1.5 (2.65)
  SBP, Week 12 | 2.0 (11.49) | -5.3 (9.45) | -2.5 (14.29) | 0.8 (6.60)
  SBP, Follow up (Week 22) | 4.0 (13.88) | -4.7 (14.50) | -2.5 (22.52) | -4.3 (3.50)
  DBP, Week 1 | -1.0 (4.08) | -3.3 (10.97) | -6.8 (6.85) | -0.5 (8.35)
  DBP, Week 2 | -1.5 (7.33) | 0.3 (1.53) | 2.0 (5.60) | -0.3 (5.44)
  DBP, Week 3 | -4.3 (6.95) | -1.0 (6.56) | -5.3 (9.57) | -4.3 (2.75)
  DBP, Week 4 | -1.0 (7.39) | -1.3 (3.79) | 1.3 (7.46) | 1.3 (6.60)
  DBP, Week 6 | -1.0 (8.04) | 7.7 (5.77) | 5.3 (11.03) | -5.5 (4.12)
  DBP, Week 8 | -2.5 (3.32) | 11.3 (7.02) | -1.5 (10.66) | -2.0 (10.39)
  DBP, Week 10 | -2.3 (3.59) | 2.7 (10.26) | -3.0 (8.83) | -4.5 (3.70)
  DBP, Week 12 | 3.5 (6.24) | -1.7 (4.73) | -3.8 (10.53) | -4.3 (6.40)
  DBP, Follow up (Week 22) | 2.8 (6.99) | -1.0 (8.72) | 3.0 (12.54) | -3.5 (5.26)

7. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: Vital sign measurements including HR was measured after 5 minutes rest before each reading. Baseline was considered as the latest pre-dose assessment. The change from Baseline is defined as the difference between the post-dose visit value and Baseline value.
Time Frame: Baseline and up to 22 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Beats per minute
  Week 1 | 0.3 (5.12) | -8.0 (3.61) | 11.5 (13.30) | -0.8 (4.27)
  Week 2 | 3.0 (11.34) | -5.3 (2.31) | 9.5 (15.15) | -5.0 (1.41)
  Week 3 | 1.3 (3.59) | -5.3 (3.79) | 10.8 (18.10) | -7.0 (5.94)
  Week 4 | 2.5 (5.45) | -5.7 (14.01) | 12.0 (15.12) | -7.8 (2.06)
  Week 6 | 7.3 (10.11) | -7.3 (6.43) | 11.0 (15.92) | -0.5 (11.50)
  Week 8 | 5.8 (8.26) | -2.7 (10.12) | 1.8 (11.30) | -11.5 (6.66)
  Week 10 | 8.3 (9.07) | 1.3 (8.02) | 0.8 (11.41) | -8.8 (10.94)
  Week 12 | -2.0 (8.68) | -10.0 (7.00) | 12.5 (11.03) | -7.8 (5.56)
  Follow up (Week 22) | -2.3 (7.14) | -6.0 (11.53) | 6.3 (20.34) | -1.3 (8.22)

8. Secondary Outcome: Change From Baseline in Body Temperature
Description: Vital sign measurements including body temperature was measured after 5 minutes rest before each reading. Baseline was considered as the latest pre-dose assessment. The change from Baseline is defined as the difference between the post-dose visit value and Baseline value.
Time Frame: Baseline and up to 22 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Celsius
  Week 1 | 0.00 (0.469) | -0.20 (0.346) | 0.18 (0.287) | 0.05 (0.265)
  Week 2 | 0.07 (0.330) | 0.03 (0.153) | -0.13 (0.250) | 0.22 (0.718)
  Week 3 | -0.10 (0.476) | -0.30 (0.265) | 0.18 (0.359) | 0.15 (0.843)
  Week 4 | -0.20 (0.327) | -0.47 (0.379) | 0.20 (0.316) | -0.15 (0.387)
  Week 6 | -0.03 (0.377) | 0.07 (0.404) | -0.10 (0.200) | -0.02 (0.457)
  Week 8 | -0.20 (0.424) | 0.03 (0.503) | -0.07 (0.377) | 0.05 (0.332)
  Week 10 | 0.00 (0.337) | 0.13 (0.252) | -0.02 (0.386) | 0.17 (0.499)
  Week 12 | -0.07 (0.427) | 0.00 (0.458) | -0.25 (0.370) | 0.02 (0.670)
  Follow up (Week 22) | -0.47 (0.862) | -0.13 (0.208) | 0.25 (0.311) | -0.18 (0.171)

9. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Vital sign measurements including respiratory rate was measured after 5 minutes rest before each reading. Baseline was considered as the latest pre-dose assessment. The change from Baseline is defined as the difference between the post-dose visit value and Baseline value.
Time Frame: Baseline and up to 22 weeks
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Breaths per minute
  Week 1 | -2.0 (1.63) | 0.7 (1.15) | -1.0 (1.41) | 0.8 (2.22)
  Week 2 | -0.5 (3.42) | 0.0 (0.00) | -1.0 (2.00) | 0.3 (1.26)
  Week 3 | 0.3 (3.10) | 1.3 (2.31) | 0.8 (0.96) | 1.5 (3.11)
  Week 4 | -2.5 (3.42) | -1.7 (2.89) | -0.5 (2.38) | 0.3 (1.71)
  Week 6 | 1.5 (5.45) | -1.0 (1.73) | -0.3 (0.96) | 2.3 (5.19)
  Week 8 | -0.3 (2.63) | 1.3 (2.31) | -1.3 (0.96) | 0.3 (1.71)
  Week 10 | 0.0 (1.63) | -0.7 (1.15) | -2.3 (1.50) | 1.0 (3.46)
  Week 12 | 1.0 (1.41) | -0.3 (2.52) | -2.5 (3.11) | 0.8 (3.59)
  Follow up (Week 22) | 0.0 (0.82) | 0.3 (3.51) | -1.5 (2.08) | 0.5 (1.00)

10. Secondary Outcome: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: 12-Lead ECGs were taken using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and corrected QT (QTc) intervals. Number of participants with any abnormal findings in ECG recordings were summarized as clinically significant and not clinically significant. Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: At Week 12
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants
  Abnormal - Not clinically significant | 1 | 1 | 1 | 0
  Abnormal - Clinically significant | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Emergent Hematology Results Relative to Normal Range
Description: Blood samples were collected to evaluate hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), erythrocytes, reticulocytes, white blood cells (WBC), total neutrophils, eosinophils, basophils, monocytes, lymphocytes, platelet count, activated partial thromboplastin time (APTT), prothrombin time (PT), fibrinogen, erythrocyte sedimentation rate (ESR). Participants were counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose lab value category was unchanged (e.g. High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if they had values that changed 'To Low' and 'To High', so the percentages may not add to 100% in such instances.
Time Frame: Up to 22 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants
  APTT, To Low | 1 | 0 | 1 | 0
  APTT, To Normal or No change | 3 | 3 | 3 | 4
  APTT, To High | 0 | 0 | 0 | 0
  Basophils, To Low | 0 | 0 | 0 | 0
  Basophils, To Normal or No change | 4 | 3 | 4 | 4
  Basophils, To High | 0 | 0 | 0 | 0
  Eosinophils, To Low | 0 | 0 | 0 | 0
  Eosinophils, To Normal or No change | 4 | 3 | 4 | 4
  Eosinophils, To High | 0 | 0 | 0 | 0
  ESR, To low | 0 | 0 | 0 | 0
  ESR, To Normal or No change | 2 | 3 | 4 | 4
  ESR, To High | 2 | 0 | 0 | 0
  Fibrinogen, To Low | 0 | 0 | 0 | 0
  Fibrinogen, To Normal or No change | 3 | 3 | 4 | 4
  Fibrinogen, To High | 1 | 0 | 0 | 0
  Hemoglobin, To Low | 1 | 1 | 2 | 0
  Hemoglobin, To Normal or No change | 3 | 2 | 2 | 4
  Hemoglobin, To High | 0 | 0 | 0 | 0
  Hematocrit, To Low | 1 | 2 | 1 | 0
  Hematocrit, To Normal or No change | 3 | 1 | 3 | 4
  Hematocrit, To High | 0 | 0 | 0 | 0
  Lymphocytes, To Low | 2 | 1 | 3 | 0
  Lymphocytes, To Normal or No change | 2 | 2 | 1 | 4
  Lymphocytes, To High | 0 | 0 | 0 | 0
  MCHC, To Low | 1 | 1 | 0 | 0
  MCHC, To Normal or No change | 3 | 2 | 4 | 4
  MCHC, To High | 0 | 0 | 0 | 0
  MCH, To Low | 1 | 0 | 0 | 0
  MCH, To Normal or No change | 3 | 3 | 4 | 4
  MCH, To High | 0 | 0 | 0 | 0
  MCV, To Low | 0 | 0 | 0 | 0
  MCV, To Normal or No change | 3 | 3 | 4 | 4
  MCV, To High | 1 | 0 | 0 | 0
  Monocytes, To Low | 1 | 0 | 0 | 0
  Monocytes, To Normal or No change | 2 | 3 | 4 | 4
  Monocytes, To High | 1 | 0 | 0 | 0
  Total neutrophils, To Low | 0 | 1 | 0 | 1
  Total neutrophils, To Normal or No change | 4 | 2 | 3 | 3
  Total neutrophils, To High | 0 | 0 | 1 | 0
  Platelet count, To Low | 0 | 0 | 0 | 0
  Platelet count, To Normal or No change | 4 | 3 | 4 | 4
  Platelet count, To High | 0 | 0 | 0 | 0
  PT, To Low | 0 | 0 | 0 | 0
  PT, To Normal or No change | 4 | 2 | 4 | 4
  PT, To High | 0 | 1 | 0 | 0
  RBC, To Low | 0 | 0 | 3 | 0
  RBC, To Normal or No change | 4 | 3 | 1 | 4
  RBC, To High | 0 | 0 | 0 | 0
  Reticulocytes, To Low | 0 | 0 | 0 | 0
  Reticulocytes, To Normal or No change | 4 | 3 | 4 | 4
  Reticulocytes, To High | 0 | 0 | 0 | 0
  WBC, To Low | 0 | 0 | 0 | 0
  WBC, To Normal or No change | 4 | 3 | 4 | 3
  WBC, To High | 0 | 0 | 0 | 1

12. Secondary Outcome: Number of Participants With Emergent Clinical Chemistry Results Relative to Normal Range
Description: Blood samples were collected to evaluate Albumin, Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Total Bilirubin, Calcium, Cholesterol, Creatine Kinase, C-Reactive protein (CRP), Creatinine, Gamma Glutamyl Transferase (GGT), Glucose, High Density Lipids (HDL), Potassium, Lactate Dehydrogenase, Low Density Lipids (LDL), Sodium, Phosphorus inorganic, Triglycerides, Total Protein and Urea. Participants were counted in the worst case category that their value changes to (low, normal or high), unless there is no change in their category. Participants whose lab value category was unchanged (e.g. High to High), or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if they had values that changed 'To Low' and 'To High', so the percentages may not add to 100% in such instances.
Time Frame: Up to 22 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants
  Albumin, To Low | 0 | 0 | 2 | 0
  Albumin, To Normal or No change | 4 | 3 | 2 | 4
  Albumin, To High | 0 | 0 | 0 | 0
  ALP, To Low | 0 | 0 | 0 | 0
  ALP, To Normal or No change | 2 | 3 | 4 | 4
  ALP, To High | 2 | 0 | 0 | 0
  ALT, To Low | 0 | 0 | 0 | 0
  ALT, To Normal or No change | 4 | 3 | 4 | 4
  ALT, To High | 0 | 0 | 0 | 0
  AST, To Low | 0 | 0 | 0 | 0
  AST, To Normal or No change | 4 | 3 | 4 | 3
  AST, To High | 0 | 0 | 0 | 1
  Total Bilirubin, To Low | 2 | 0 | 0 | 0
  Total Bilirubin, To Normal or No change | 2 | 3 | 4 | 4
  Total Bilirubin, To High | 0 | 0 | 0 | 0
  Calcium, To Low | 1 | 0 | 1 | 1
  Calcium, To Normal or No change | 3 | 3 | 3 | 3
  Calcium, To High | 0 | 0 | 0 | 0
  Cholesterol, To Low | 0 | 0 | 0 | 0
  Cholesterol, To Normal or No change | 2 | 2 | 4 | 4
  Cholesterol, To High | 2 | 1 | 0 | 0
  Creatine Kinase, To Low | 0 | 1 | 0 | 0
  Creatine Kinase, To Normal or No change | 3 | 2 | 4 | 3
  Creatine Kinase, To High | 1 | 0 | 0 | 1
  CRP, To Low | 0 | 0 | 0 | 0
  CRP, To Normal or No change | 2 | 3 | 4 | 4
  CRP, To High | 2 | 0 | 0 | 0
  Creatinine, To Low | 0 | 1 | 1 | 0
  Creatinine, To Normal or No change | 4 | 2 | 3 | 4
  Creatinine, To High | 0 | 0 | 0 | 0
  GGT, To Low | 0 | 0 | 0 | 0
  GGT, To Normal or No change | 4 | 3 | 4 | 4
  GGT, To High | 0 | 0 | 0 | 0
  Glucose, To Low | 0 | 0 | 0 | 1
  Glucose, To Normal or No change | 1 | 2 | 3 | 2
  Glucose, To High | 3 | 1 | 1 | 1
  HDL, To Low | 0 | 1 | 0 | 0
  HDL, To Normal or No change | 4 | 2 | 4 | 4
  HDL, To High | 0 | 0 | 0 | 0
  Potassium To Low | 2 | 1 | 1 | 0
  Potassium, To Normal or No change | 2 | 2 | 3 | 4
  Potassium, To High | 0 | 0 | 0 | 0
  Lactate Dehydrogenase, To Low | 0 | 0 | 0 | 0
  Lactate Dehydrogenase, To Normal or No change | 3 | 3 | 3 | 3
  Lactate Dehydrogenase, To High | 1 | 0 | 1 | 1
  LDL, To Low | 0 | 0 | 0 | 0
  LDL, To Normal or No change | 2 | 2 | 4 | 4
  LDL, To High | 2 | 1 | 0 | 0
  Sodium, To Low | 0 | 0 | 0 | 0
  Sodium, To Normal or No change | 4 | 3 | 4 | 4
  Sodium, To High | 0 | 0 | 0 | 0
  Phosphorus inorganic, To Low | 0 | 0 | 0 | 0
  Phosphorus inorganic, To Normal or No change | 4 | 3 | 4 | 4
  Phosphorus inorganic, To High | 0 | 0 | 0 | 0
  Triglycerides, To Low | 0 | 0 | 0 | 1
  Triglycerides, To Normal or No change | 4 | 3 | 4 | 3
  Triglycerides, To High | 0 | 0 | 0 | 0
  Total Protein, To Low | 1 | 1 | 1 | 0
  Total Protein, To Normal or No change | 3 | 2 | 3 | 4
  Total Protein, To High | 0 | 0 | 0 | 0
  Urea, To Low | 1 | 0 | 0 | 1
  Urea, To Normal or No change | 3 | 3 | 3 | 3
  Urea, To High | 0 | 0 | 1 | 0

13. Secondary Outcome: Number of Participants With Urinalysis Dipstick Findings
Description: Urine samples were collected for analysis of presence of glucose and protein in urine by dipstick method. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine protein and glucose can be read as negative, Trace, 1+, 2+ and 3+, indicating proportional concentrations in the urine sample
Time Frame: Up to 22 weeks
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants
  Week 4, Glucose, 1+ | 0 | 0 | 0 | 0
  Week 4, Glucose, 2+ | 0 | 0 | 0 | 0
  Week 4, Glucose, 3+ | 0 | 0 | 0 | 1
  Week 4, Glucose, Negative | 4 | 3 | 4 | 3
  Week 4, Glucose, Trace | 0 | 0 | 0 | 0
  Week 4, Protein, 1+ | 1 | 0 | 1 | 0
  Week 4, Protein, 2+ | 0 | 0 | 0 | 0
  Week 4, Protein, 3+ | 0 | 0 | 0 | 0
  Week 4, Protein, Negative | 1 | 3 | 2 | 4
  Week 4, Protein, Trace | 2 | 0 | 1 | 0
  Week 8, Glucose, 1+ | 0 | 0 | 0 | 1
  Week 8, Glucose, 2+ | 0 | 0 | 0 | 0
  Week 8, Glucose, 3+ | 0 | 0 | 0 | 0
  Week 8, Glucose, Negative | 4 | 3 | 4 | 3
  Week 8, Glucose, Trace | 0 | 0 | 0 | 0
  Week 8, Protein, 1+ | 0 | 0 | 1 | 0
  Week 8, Protein, 2+ | 0 | 0 | 0 | 0
  Week 8, Protein, 3+ | 0 | 0 | 0 | 0
  Week 8, Protein, Negative | 1 | 3 | 3 | 2
  Week 8, Protein, Trace | 3 | 0 | 0 | 2
  Week 12, Glucose, 1+ | 0 | 0 | 0 | 0
  Week 12, Glucose, 2+ | 0 | 0 | 0 | 0
  Week 12, Glucose, 3+ | 0 | 0 | 0 | 0
  Week 12, Glucose, Negative | 4 | 3 | 4 | 4
  Week 12, Glucose, Trace | 0 | 0 | 0 | 0
  Week 12, Protein, 1+ | 0 | 0 | 0 | 1
  Week 12, Protein, 2+ | 0 | 0 | 0 | 0
  Week 12, Protein, 3+ | 0 | 0 | 0 | 0
  Week 12, Protein, Negative | 3 | 3 | 3 | 3
  Week 12, Protein, Trace | 1 | 0 | 1 | 0
  Follow up (Week 22), Glucose, 1+ | 0 | 0 | 0 | 0
  Follow up (Week 22), Glucose, 2+ | 0 | 0 | 0 | 0
  Follow up (Week 22), Glucose, 3+ | 0 | 0 | 0 | 0
  Follow up (Week 22), Glucose, Negative | 4 | 3 | 4 | 4
  Follow up (Week 22), Glucose, Trace | 0 | 0 | 0 | 0
  Follow up (Week 22), Protein, 1+ | 1 | 0 | 1 | 0
  Follow up (Week 22), Protein, 2+ | 0 | 0 | 0 | 0
  Follow up (Week 22), Protein, 3+ | 0 | 0 | 0 | 0
  Follow up (Week 22), Protein, Negative | 2 | 3 | 3 | 3
  Follow up (Week 22), Protein, Trace | 1 | 0 | 0 | 1

14. Secondary Outcome: Number of Participants With Anti-GSK3196165 Antibody Test Results
Description: Serum samples were collected and tested for presence of antibodies that bind to GSK3196165. The presence of treatment emergent anti-drug antibodies (ADA) were determined using a GSK3196165 bridging style ADA assay with a bio-analytically determined cut point determined during assay validation. Samples taken after dosing with GSK3196165 that have a value at or above the cut-point were considered treatment-emergent ADA-positive. These ADA positive samples were further evaluated in a confirmatory assay, and confirmed positive samples were further characterized by assessment of titer. Baseline was considered as the latest pre-dose assessment. Number of participants with post-Baseline negative or positive anti-GSK3196165 antibody test results were presented.
Time Frame: Weeks 2, 4, 12 and 22
Population: Immunogenicity Population. The immunogenicity Population included all participants in the ITT Population, who had at least one immunogenicity assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Participants
  Week 2, Positive | 0 | 0 | 0 | 0
  Week 2, Negative | 4 | 3 | 4 | 4
  Week 4, Positive | 0 | 0 | 0 | 0
  Week 4, Negative | 4 | 3 | 4 | 4
  Week 12, Positive | 0 | 0 | 0 | 0
  Week 12, Negative | 4 | 3 | 4 | 4
  Week 22 (Follow up), Positive | 0 | 0 | 0 | 0
  Week 22 (Follow up), Negative | 4 | 3 | 4 | 4

15. Secondary Outcome: Change From Baseline in Disease Activity Score for 28 Different Joints C-reactive Protein (DAS28 [CRP]) at All Indicated Timepoints
Description: DAS28 (CRP) is a measure of disease activity in rheumatoid arthritis obtained by examination of 28 joints for swelling and tenderness using CRP as a blood biomarker for inflammation. Its components include: Tender/Painful Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), CRP and Patient's Global Assessment of Arthritis. DAS28 (CRP) was calculated by 0.56 (square root of TJC28)+ 0.28 (square root of SJC28)+ 0.36 (natural logarithm [CRP+1])+ (0.014*patients global assessment)+0.96. Scores ranges from 0 to infinity, where higher scores indicates high disease activity. Scores higher than 5.1 indicates high disease activity and scores lower than 2.6 indicates remission. Baseline was considered as the latest pre-dose assessment. The change from Baseline is defined as the difference between the post-dose visit value and Baseline value. Adjusted mean and standard error of adjusted mean are presented using Mixed Model for Repeated Measures.
Time Frame: Baseline, up to Week 22
Population: ITT Population
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4
Scores on a scale
  Week 1 | -0.2179 (0.44925) | -1.3289 (0.51977) | -0.7356 (0.42589) | -0.7511 (0.42569)
  Week 2 | 0.1643 (0.48797) | -0.9744 (0.56457) | -0.7262 (0.46260) | -0.6404 (0.46238)
  Week 4 | -0.0887 (0.59912) | -1.5462 (0.69316) | -0.9781 (0.56796) | -1.2502 (0.56769)
  Week 6 | -0.5455 (0.55367) | -0.8664 (0.64058) | -0.7330 (0.52487) | -1.0048 (0.52463)
  Week 8 | -0.2710 (0.69364) | -0.9231 (0.80253) | -0.8209 (0.65757) | -1.2375 (0.65726)
  Week 12 | -0.8234 (0.76338) | -1.1810 (0.88321) | -0.6383 (0.72368) | -0.9415 (0.72335)
  Week 22 (Follow-up) | -0.3044 (0.62302) | -1.7320 (0.72082) | 0.2371 (0.59062) | -1.0976 (0.59035)
Statistical Analysis 1: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -1.1110, 95% CI 2-sided [-2.7186 to 0.4965] — Week 1. The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 2: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = -0.5177, 95% CI 2-sided [-1.9040 to 0.8685] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -0.5332, 95% CI 2-sided [-1.9140 to 0.8475] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -1.1387, 95% CI 2-sided [-2.8848 to 0.6075] — Week 2. The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 5: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = -0.8905, 95% CI 2-sided [-2.3962 to 0.6153] — [estimate comment as in outcome 15, analysis 4]
Statistical Analysis 6: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -0.8047, 95% CI 2-sided [-2.3045 to 0.6951] — [estimate comment as in outcome 15, analysis 4]
Statistical Analysis 7: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -1.4575, 95% CI 2-sided [-3.6013 to 0.6863] — Week 4. The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 8: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = -0.8894, 95% CI 2-sided [-2.7381 to 0.9593] — [estimate comment as in outcome 15, analysis 7]
Statistical Analysis 9: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -1.1615, 95% CI 2-sided [-3.0028 to 0.6799] — [estimate comment as in outcome 15, analysis 7]
Statistical Analysis 10: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -0.3209, 95% CI 2-sided [-2.3021 to 1.6603] — Week 6. The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 11: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = -0.1876, 95% CI 2-sided [-1.8960 to 1.5209] — [estimate comment as in outcome 15, analysis 10]
Statistical Analysis 12: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -0.4593, 95% CI 2-sided [-2.1610 to 1.2424] — [estimate comment as in outcome 15, analysis 10]
Statistical Analysis 13: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -0.6521, 95% CI 2-sided [-3.1342 to 1.8300] — Week 8. The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 14: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = -0.5499, 95% CI 2-sided [-2.6903 to 1.5904] — [estimate comment as in outcome 15, analysis 13]
Statistical Analysis 15: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -0.9665, 95% CI 2-sided [-3.0984 to 1.1654] — [estimate comment as in outcome 15, analysis 13]
Statistical Analysis 16: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -0.3576, 95% CI 2-sided [-3.0892 to 2.3740] — Week 12. The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 17: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = 0.1851, 95% CI 2-sided [-2.1704 to 2.5407] — [estimate comment as in outcome 15, analysis 16]
Statistical Analysis 18: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -0.1181, 95% CI 2-sided [-2.4643 to 2.2281] — [estimate comment as in outcome 15, analysis 16]
Statistical Analysis 19: Comparison: Placebo vs GSK3196165 45 mg; Test type: Other; Mean Difference (Net) = -1.4276, 95% CI 2-sided [-3.6569 to 0.8018] — Week 22 (Follow up). The analysis method was mixed-model for repeated measures with Visit,Treatment group,Visit by Treatment interaction,Baseline DAS28(CRP),and Visit by Baseline DAS28(CRP) interaction as fixed effects
Statistical Analysis 20: Comparison: Placebo vs GSK3196165 90 mg; Test type: Other; Mean Difference (Net) = 0.5415, 95% CI 2-sided [-1.3810 to 2.4639] — [estimate comment as in outcome 15, analysis 19]
Statistical Analysis 21: Comparison: Placebo vs GSK3196165 180 mg; Test type: Other; Mean Difference (Net) = -0.7932, 95% CI 2-sided [-2.7080 to 1.1217] — [estimate comment as in outcome 15, analysis 19]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (non-serious AEs) were collected from the start of the study treatment up to Week 22.
Description: SAEs and non-serious AEs were reported for the ITT Population.
Arm/Group | Placebo | GSK3196165 45 mg | GSK3196165 90 mg | GSK3196165 180 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 3/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | GSK3196165 45 mg (N=3) | GSK3196165 90 mg (N=4) | GSK3196165 180 mg (N=4)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | GSK3196165 45 mg (N=3) | GSK3196165 90 mg (N=4) | GSK3196165 180 mg (N=4)
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT03028467/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/67/NCT03028467/SAP_001.pdf